CLINICAL TRIAL: NCT01810081
Title: Study of Relationship Between Gallstones and Concomitant Gastric Helicobacter Pylori Infection
Brief Title: Gallstones and Concomitant Gastric Helicobacter Pylori Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, M.Umit UGURLU, Assist.Prof., Marmara University
Other Study IDs: B.30.2.MAR.0.01.02/AEK/73
Record Dates: First submitted 2013-03-06; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Cholelithiasis
Keywords: Cholelithiasis; Gastric H.Pylori infection; H.Pylori infection; Gastric mucosa
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cholecystectomy: cholecystectomy group: H.Pylori infection in gall bladder

SUMMARY:
In this study, the presence of H.Pylori in the gallbladder mucosa of patients with symptomatic gallstones undergoing cholecystectomy was investigated. Concomitant H.Pylori infection of the gastric mucosa was also investigated to study the relationship of gastric H.Pylori infection to gallstones. It was hypothesized that H.Pylori infection of the gastric mucosa may have a role in the formation of gallstones.

DETAILED DESCRIPTION:
Gallstone disease is one of the most common problems affecting the digestive tract where autopsy reports show a prevalence of 11-36% . The prevalence of gallstones is related to many factors including age, gender, and ethnic background. Women are three times more likely to develop gallstones than man and first-degree relatives have a two-fold increased prevalence . However, the etiology of gallstone formation beginning with the change in the composition of bile, leading to stones is not clear.

The association between Helicobacter pylori (H.Pylori) and gallstones has been investigated but not clearly demonstrated. H.Pylori is a gram negative and micro-aerophilic microorganism that can cause chronic gastritis, gastric and duodenal ulcers, gastric adenocarcinoma and lymphoma of gastric mucosa-related lymphoid tissue (MALToma) . Relationship of H.Pylori with diseases of organs other than the stomach and duodenum has also been investigated and reported . H.Pylori have been detected in the gallbladder mucosa of patients with gallstones .

In this study, the presence of H.Pylori in the gallbladder mucosa of patients with symptomatic gallstones undergoing cholecystectomy was investigated. Concomitant H.Pylori infection of the gastric mucosa was also investigated to study the relationship of gastric H.Pylori infection to gallstones. It was hypothesized that H.Pylori infection of the gastric mucosa may have a role in the formation of gallstones.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cholecystitis, cholangitis, biliary and hepatic tumors, Crohn's disease, and previous gastric surgery were not considered suitable for evaluation.

Exclusion Criteria:

* Patients undergoing ERCP (endoscopic retrograde cholangio-pancreatography) and patients who have received H.Pylori eradication treatment in the last 6 month were also excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ninety-four patients with symptomatic gallstones undergoing laparoscopic cholecystectomy were enrolled for the study.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Gallstones and concomitant H.Pylori infection of the gastric mucosa | 3 months
  The relationship between gastric H.Pylori infection and comcomitant gallstones will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: A.Ozdemir Aktan, md,PROF, Study Director — Marmara University
Locations (1):
- marmara University School of Medicine, Istanbul, Turkey (Türkiye)